CLINICAL TRIAL: NCT05009290
Title: A Phase III Randomized, Placebo-Controlled, Double-Blind Study of SHR3680 Plus Androgen Deprivation Therapy (ADT) Versus ADT in Patients With High-Risk Localized or Locally Advanced Prostate Cancer Undergoing Radical Prostatectomy
Brief Title: A Trial of SHR3680 in Prostate Cancer Patients Who Are Candidates for Radical Prostatectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3680-III-302
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-08

CONDITIONS: Patients With High-risk Localized or Locally Advanced Prostate Cancer Who Are Candidates for Radical Prostatectomy

STUDY DESIGN:
Intervention Model Description: SHR3680 + ADT compared with placebo + ADT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group：SHR3680 + ADT (Experimental)
  Interventions: Drug: SHR3680
- Treatment group : Placebo + ADT (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR3680 — Treatment group: SHR3680 240 mg orally once daily before or after breakfast, 28 days per cycle for a total of 12 treatment cycles (6 cycles before and 6 cycles following radical prostatectomy).
  Goserelin acetate sustained-release depot: 10.8 mg administered subcutaneously into the anterior abdominal wall once every 3 cycles (12 weeks) for a total of 12 cycles.
  Arms: Treatment group：SHR3680 + ADT
Drug: Placebo — Treatment group ：Placebo 240 mg orally once daily before or after breakfast, 28 days per cycle for a total of 12 treatment cycles (6 cycles before and 6 cycles following radical prostatectomy).
  Goserelin acetate sustained-release depot: 10.8 mg administered subcutaneously into the anterior abdominal wall once every 3 cycles (12 weeks) for a total of 12 cycles.
  Arms: Treatment group : Placebo + ADT

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR3680 plus androgen deprivation therapy (ADT) vs. placebo plus ADT in patients with high-risk localized or locally advanced prostate cancer using pathologic complete response (pCR) rate and metastasis-free survival (MFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 18 years old;
2. ECOG PS score of 0 or 1;
3. Pathologically diagnosed as prostate adenocarcinoma;
4. High-risk patients
5. No distant metastasis (clinical staging of M0) as determined by BICR of imaging examinations;
6. Subjects who are candidates for and plan to undergo radical prostatectomy (removal of the entire prostate and seminal vesicle plus pelvic lymphadenectomy);

Exclusion Criteria:

1. Subjects who received any prior treatment for prostate cancer, except medical ADT and/or first-generation androgen receptor antagonists (such as bicalutamide) for not more than 4 weeks;
2. Subjects who received any other investigational products or underwent major surgery within 4 weeks prior to randomization;
3. Subjects who are planning bilateral orchidectomy during the treatment period of the study;
4. Subjects with dysphagia, chronic diarrhea, intestinal obstruction, or other factors affecting drug intake and absorption;
5. Subjects with a history of epilepsy, or diseases that can induce seizures occurred within 12 months prior to randomization (including a history of transient ischemic attack, stroke, traumatic brain injury, and cognitive impairment, requiring hospitalization);
6. Subjects with active heart disease within 6 months prior to randomization, including: severe/unstable angina pectoris, myocardial infarction, symptomatic congestive heart failure, and ventricular arrhythmias requiring medical treatment;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1256 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2031-10-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate (assessed by pathology BICR) | 36 months since the first subject will be enrolled.
  Defined as the proportion of subjects with no residual tumor detected in prostatectomy specimens by H&E staining and ancillary immunohistochemistry (if necessary) as assessed by pathology BICR.
MFS (assessed by imaging BICR). | 84 months since the first subject will be enrolled.
  Defined as the time from the date of randomization to the date of first occurrence of BICR-confirmed radiographic distant metastasis, accidental pathologic finding of distant metastasis, or death from any cause (whichever occurs first), regardless of whether the subject reveives any other anti-tumor therapy or has missing (or unevaluable) tumor assessments.

SECONDARY OUTCOMES:
MFS (investigator-assessed). | 84 months since the first subject will be enrolled.
  Defined as the time from the date of randomization to the date of first occurrence of investigator-assessed radiographic distant metastasis to the bone or soft tissue, accidental pathologic finding of distant metastasis, or death from any cause (whichever occurs first), regardless of subsequent anti-tumor treatment or missing (or unevaluable) tumor assessments.
PSA response rate. | 25 months since the first subject will be enrolled.
  Defined as the proportion of subjects with a ≥ 90% decrease in PSA levels from baseline on Day 1 of Cycle 4.
PSM rate. | 31 months since the first subject will be enrolled.
  Defined as the proportion of subjects without tumor cells detected in the margin of prostatectomy pathological specimens following H&E staining and ancillary immunohistochemistry (if necessary), as assessed by local pathologists.
Time to BCR. | 42 months since the first subject will be enrolled.
  Defined as the time from the date of randomization to the time of BCR (i.e. two consecutive PSA rise ≥ 0.2 ng/mL following radical prostatectomy).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality, China